CLINICAL TRIAL: NCT03654430
Title: Longitudinal Study by 2D-speckle-tracking Echocardiography of the Ventricular Wall Motion During Postnatal Adaptation
Brief Title: Study by 2D-strain of the Ventricular Wall Motion During Postnatal Adaptation
Acronym: BABYSTRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC18.014
Record Dates: First submitted 2018-05-14; First posted 2018-08-31 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Healthy
Keywords: Left ventricular Twist; 2D-speckle-tracking; Postnatal adaptation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Newborns (Other)
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Two echocardiographies will be performed in healthy newborns: The first between day 2 and day 5 of life, the second between day 60 and day 90 of life

SUMMARY:
The left ventricular torsion during systole and diastole is a normal dynamic mechanism which participates in the ejection and the filling of the left ventricle. Postnatal hemodynamic modifications are major and probably affect this mechanism. The aim of this study is to compare the left ventricular twist in healthy newborns, between their first days of life and their third month of life, using the 2D-speckle tracking echocardiography.

DETAILED DESCRIPTION:
The left ventricular torsion during systole and diastole is a normal dynamic mechanism which participates in the ejection and the filling of the left ventricle. Postnatal hemodynamic modifications are major and probably affect this mechanism.

The main objective is to compare the left ventricular twist mechanism in healthy newborns, at birth and at their third month of life, using the peak LV twist as primary endpoint. Secondarily, we compare other LV rotation and deformation parameters during the same period: peak LV torsion, peak LV twist rate, peak LV untwist rate, circumferential strain and radial strain. Finally, we compare the endo- and epicardial LV deformation, using the inner and outer circumferential strain as endpoints.

This is a longitudinal, prospective and monocentric study in the Grenoble-Alpes University Hospital between April 2018 and September 2018.

The number of required subjects is 30 with a statistical power of 80% and a p-value of 0,05

ELIGIBILITY:
Inclusion Criteria:

* Newborn hospitalized in the Grenoble University Hospital Maternity Unit
* Aged between 2 and 5 day of life at the first echocardiography
* Social security affiliation
* Signature of the consent document by both parents

Exclusion Criteria:

* Birth before 37 weeks gestation
* Birth weight < 2,5kg or > 4,5kg
* Gestational Diabetes Mellitus during pregnancy
* Fetal heart disease

Ages: 2 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Left ventricular Twist | 3 months
  Peak LV twist (°)

SECONDARY OUTCOMES:
Left ventricular Rotation | 3 months
  Basal Rotation (°); Apical Rotation (°); Peak LV twist rate (°/s); Peak LV systolic torsion
Untwist | 3 months
  Peak LV Untwist rate (°/sec)
Left ventricular deformation | 3 months
  Basal and Apical Circumferential Strain (%); Basal and Apical Radial Strain (%)
Comparison between Endocardial and Epicardial deformation | 3 months
  Inner and Outer Circumferential Strain (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Johanne Auriau, Grenoble, France